CLINICAL TRIAL: NCT03797027
Title: Effects of Abdominal Cushion on Percutaneous Nephrostolithotomy in Prone Position: a Randomized Controlled Trial
Brief Title: Effects of Abdominal Cushion on PCNL in Prone Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice president, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Honglin Sun
Record Dates: First submitted 2019-01-05; First posted 2019-01-08 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Kidney Stone
Keywords: Percutaneous nephrolithotomy; cushion
MeSH Terms: conditions — Kidney Calculi | interventions — Nephrolithotomy, Percutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No cushion (Other): Patients in no cushion group undergo prone percutaneous nephrolithotomy without an abdominal cushion
  Interventions: Device: Percutaneous Nephrolithotomy without an abdominal cushion
- 5 cm cushion (Other): Patients in 5 cm cushion group undergo prone percutaneous nephrolithotomy with an 5 cm abdominal cushion
  Interventions: Device: Percutaneous Nephrolithotomy with an 5 cm abdominal cushion
- 10 cm cushion (Other): Patients in 10 cm cushion group undergo prone percutaneous nephrolithotomy with an 10 cm abdominal cushion
  Interventions: Device: Percutaneous Nephrolithotomy with an 5 cm abdominal cushion

INTERVENTIONS:
Device: Percutaneous Nephrolithotomy without an abdominal cushion — patients undergo prone PNCL without an abdominal cushion
  Arms: No cushion
Device: Percutaneous Nephrolithotomy with an 5 cm abdominal cushion — patients undergo prone PNCL with an 5 cm abdominal cushion
  Arms: 5 cm cushion
Device: Percutaneous Nephrolithotomy with an 5 cm abdominal cushion — patients undergo prone PNCL with an 10 cm abdominal cushion
  Arms: 10 cm cushion

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is the first choice for the treatment of ≥ 2cm renal stones. The positions of PCNL includes supine, prone and lateral. PCNL has been performed in my center for nearly twenty years. The prone position is routinely used. Generally speaking, an abdominal cushion is used to raise the abdominal in the prone position, in order to provide an adequate exposure of kidney, increase the intercostal space, decrease the mobility of kidney and lower the risk of pleura injury. However, there is no consensus and criterion on the height of abdominal cushion. With largely increased PCNL procedures and various BMI, precise evaluation of abdominal cushion is needed. In the preliminary work, the investigators measured the sunken height of waist of 100 patients in the prone position without a abdominal cushion. The results showed that the mean BMI of 100 patients was 23.45 (16.79-36.98) and the range of sunken height of waist was 2-7 cm. Therefore, the investigators are planning to conduct a randomized controlled study to compare the safety and efficacy among no cushion group, 5 cm cushion group and 10 cm cushion group. To clarify the relationship between height of abdominal cushion and BMI, the nurse could prepare the appropriate cushion the day before surgery, which would decrease operating time and accelerate postoperative recovery.

DETAILED DESCRIPTION:
1. Background Percutaneous nephrolithotomy (PCNL) is the first choice for the treatment of ≥ 2cm renal stones.The positions of PCNL includes supine, prone and lateral. PCNL has been performed in my center for nearly twenty years. The prone position is routinely used. Generally speaking, an abdominal cushion is used to raise the abdominal in the prone position, in order to provide an adequate exposure of kidney, increase the intercostal space, decrease the mobility of kidney and lower the risk of pleura injury. However, there is no consensus and criterion on the height of abdominal cushion. With largely increased PCNL procedures and various BMI, precise evaluation of abdominal cushion is needed. In the preliminary work, the investigators measured the sunken height of waist of 100 patients in the prone position without a abdominal cushion. The results showed that the mean BMI of 100 patients was 23.45 (16.79-36.98) and the range of sunken height of waist was 2-7 cm. Therefore, the investigators are planning to conduct a randomized controlled study to compare the safety and efficacy among no cushion group, 5 cm cushion group and 10 cm cushion group. To clarify the relationship between height of abdominal cushion and BMI, the nurse could prepare the appropriate cushion the day before surgery, which would decrease operating time and accelerate postoperative recovery.
2. Purpose To investigate effects of different height of abdominal cushion on prone PCNL, in terms of intraoperative parameters. Our study could provide high quality of evidences on making criteria of perioperative nurse.
3. Design 3.1 Participant： A single randomized controlled study 3.2 Number of cases： 180 patients who are candidates for PCNL will be enrolled in this study. By 1:2 simple random sampling technique, patients will be assigned to 60-patient no cushion PCNL and 120-patient cushion PCNL (60-patient for 5 cm cushion and 60-patient for 10 cm cushion).

   *(Assuming SFR (1 month after procedure) with cushion PCNL of 90% and expected rate of 70% with no cushion PCNL, the sample size for each group are calculated as 120 and 60 [power > 0.90 with a type I error rate < 0.05.]
4. Candidate:

   4.1 Included criterion：
   * Willing to receive PCNL
   * Aged 18-70 years
   * Normal renal function
   * ASA scoreⅠ to Ⅱ 4.2 Excluded criterion：
   * Uncorrected coagulopathy and active urinary tract infection (UTI)
   * Patients who underwent transplant or urinary diversion.
   * Congenital abnormalities. 4.3 Excluded from the study after inclusion Patients will be excluded from the study if the undergoing standard PNL/mini-perc have purulent fluid in the initial puncture.

   Patients with positive preoperative urine culture should be treated with suitable antibiotics based on the culture sensitivity result for at least 72 h before PCNL. Patients who have negative urine culture should receive a single dose of broad spectrum antibiotic prophylaxis just prior to the procedure. Patients who are going to receive PCNL would get a envelope including a randomized number and consent letter.
5. Surgical technique

   Under general anaesthesia, each patient is initially placed in the lithotomy position, and a 5 Fr or 6Fr ureteral catheter is inserted to the kidney and fixed with a 16 Fr Foley catheter. Then the patient is turned to the prone position. An abdominal cushion is used according to the randomized number. The choice of using C-arm fluoroscopic or ultrasonography guidance or a combination fashion for the percutaneous access was made at the discretion of the treating urologist. The length of the needle from skin to the collecting system is measured to ensure that the length of dilator is appropriate. No patient underwent bilateral simultaneous PCNL and patients with bilateral stones underwent surgery 4 weeks apart. The access tract is dilated with a fascial dilator from 8F up to 18F. The investigators defined access to the collecting system as gaining entry to the targeted urinary system and desired calix. For some complex cases, when indicated requiring multiple tracts, additional tracts were created in the same session. The stone was fragmented by pneumatic lithotripsy or Holmium:YAG laser lithotripsy through 8/9.8F semirigid ureteroscope (Richard Wolf, Germany). The large fragments were extracted with a forceps and small fragments were flushed out with an endoscopic pulsed perfusion pump. A silastic nephrostomy tube was placed at the end of procedure and a 4-6Fr double pigtail ureteral stent was left for 2 weeks after operation. X-ray check for residual stone fragments is also performed at the end of the procedure.

   Patients were candidates for the tubeless procedure only when the following strict conditions were met: single percutaneous tract, absence of major perforation of collecting system and bleeding, complete stone clearance assessed by intraoperative nephroscopy and fluoroscopy at the end of the procedure. For a tubeless procedure, the flank was compressed for 5 min. Patient was monitored for postoperative complications.
6. Data collection

Data for the 2 groups -demographic characteristics, time of puncture and dilation, site of target calix, site of access, S.T.O.N.E score, hemoglobin drop, postoperative pain, duration of procedure, hospital stay, cases of tubeless, complications (modified Clavin system), stone clearance (SFR of postoperative day 1 and 1 month follow-up) and the need for auxiliary treatment (for example, re-PCNL, RIRS and ESWL) - are compared.

ELIGIBILITY:
Inclusion Criteria:

* Willing to receive PCNL
* Aged 18-70 years
* Normal renal function
* ASA scoreⅠ to Ⅱ

Exclusion Criteria:

* Uncorrected coagulopathy and active urinary tract infection (UTI)
* Patients who underwent transplant or urinary diversion.
* Congenital abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
time of puncture and dilation | intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D & MD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China